CLINICAL TRIAL: NCT05816694
Title: The Efficacy and Safety of Nanoparticle Albumin-bound (NAB)-Paclitaxel Plus Cisolation Versus CEP (Cisplatin, Epirubicin,Cyclophosphamide) in Induction Therapy for Thymoma: a Study for a Single-center Prospective Phase II Randomized Controlled Train.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peng Liu (Other)
Responsible Party: Sponsor-Investigator, Peng Liu, Director, Shanghai Zhongshan Hospital
Organization: Shanghai Zhongshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2021-584R2
Record Dates: First submitted 2023-03-27; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Histological or Cytological Confirmed Stage Ⅲ and Ⅳa Thymoma
Keywords: nanoparticle albumin-bound (NAB)-paclitaxel plus Cisolation; CEP (cisplatin, epirubicin,cyclophosphamide); thymoma
MeSH Terms: conditions — Thymoma | interventions — 130-nm albumin-bound paclitaxel; Cisplatin; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CEP (Active Comparator): Cisplatin was administered as 50 mg/m2 IV infusion on Day 1; Epirubicin was administered as 75 mg/m2 IV infusion on Day 1; Cyclophosphamide was administered as 500 mg/m2IV infusion on Day 1 of each 3-week cycle.Patients will receive maximum of 4 cycles if they do not meet the criteria for removal from the study.
  Interventions: Drug: Cisplatin plus Epirubicin plus Cyclophosphamide
- NAB-Paclitaxel (Experimental): NAB-Paclitaxel will be administered as 125 mg/m2 IV infusion on Day 1 、Day8 of each 3-week cycle. Cisplatin will be administered as 75 mg/m2 IV infusion on Day 1 of each 3-week cycle. Patients will receive maximum of 4 cycles if they do not meet the criteria for removal from the study.
  Interventions: Drug: NAB-Paclitaxel plus Cisplatin

INTERVENTIONS:
Drug: NAB-Paclitaxel plus Cisplatin — NAB-Paclitaxel will be administered as 125 mg/m2 IV infusion on Day 1 、Day8 of each 3-week cycle. Cisplatin will be administered as 75 mg/m2 IV infusion on Day 1 of each 3-week cycle. Patients will receive maximum of 4 cycles if they do not meet the criteria for removal from the study.
  Arms: NAB-Paclitaxel
Drug: Cisplatin plus Epirubicin plus Cyclophosphamide — Cisplatin was administered as 50 mg/m2 IV infusion on Day 1; Epirubicin was administered as 75 mg/m2 IV infusion on Day 1; Cyclophosphamide was administered as 500 mg/m2IV infusion on Day 1 of each 3-week cycle.Patients will receive maximum of 4 cycles if they do not meet the criteria for removal from the study.
  Arms: CEP

SUMMARY:
This study for a single-center prospective phase II randomized controlled train to assess the efficacy and safety of Induction therapy on thymoma .Methods patients with thymoma (stage Ⅲ and stage Ⅳa) were treated with 2 cycles of (NAB)-paclitaxel plus Cisolation (Paclitaxel For Injection(Aalbumin Bound）125 mg/m2 Day 1 、Day8 ,Cisplatin 75 mg/m2 Day 1of each 3-week cycle）or CEP(cisplatin 50 mg/m2 Day 1, epirubicin 75 mg/m2 Day 1,cyclophosphamide 500 mg/m2 Day 1 of each 3-week cycle). Following chemotherapy to evaluate the patient for operation. Patients without undergo surgery will be continued to receive 2 cycles of Primary chemotherap.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years；
* Histological or cytological confirmed stage Ⅲ and Ⅳa thymoma;
* PET/CT or CT/MRI with at least one objectively measurable or evaluable lesion；
* Life expectancy >12months；
* ECOG PS 0-1；

  --Patients with thymoma metastasis；
* No found the other malignant tumors (expect has been controlled Carcinoma in situ of the cervix and Basal Cell Carcinoma）；
* Informed consent was signed before the study began；
* Normal Bone marrow hematopoiesis and renal function，Blood routine: absolute neutrophil count≥1,500/uL，Hb>8.0g/dL，PLT>80×10*9/L，AST≤ 1.5 times the upper limit of normal，TBIL ≤1.5 times the upper limit of normal，calculated creatinine clearance ≤110µmol/L，blood urea nitrogen≤7.1mmol/L；
* Cardiac function: LVEF≥55%；
* Patients who have not active bleeding or coagulopathy before enrollment；

Exclusion Criteria:

* -Patients who have been found thymoma metastasis；
* Patients with uncontrolled lung disease, Serious infection,active peptic ulcers, coagulation diaorders, Uncontrolled severe diabetes, connective tissue diseases or Bone marrow suppression and Induction therapy for intolerance；
* Peripheral neuropathy ≥ Grade 2 (NCI-CTCAE version 5.0 )；
* Significant organ dysfunction: such as respiratory failure, NYHA classification Class III or IV, chronic congestive heart failure, decompensation Hepatic or renal insufficiency, high blood pressure（SBP> 180 mmHg or DBP> 100mmHg）；
* Pregnant and lactating women；
* patients without undergo preoperative puncture biopsy or induction therapy；
* Patients with active uncontrollable neurological, mental disease or mental disorder, poor compliance, unable to cooperate and describe the treatment response；
* Patients who have received any other investigational drug treatment or participated in any other clinical trials within 30 days prior to enrollment in this study；
* Known HIV infection or active infection with HBV, HCV. Patients who are infected with HBV but not active hepatitis at the same time are not excluded；
* Patients with uncontrollable Stable myasthenia gravis or uncontrollable Serious autoimmune disease such as fulminant DIC；
* Patients who are known to be allergic or intolerant to chemotherapy drugs；
* severe-trauma；
* Patients who have received any other investigational drug treatment or participated in any other clinical trials within 30 days prior to enrollment in this study；

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-30 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
overall response rate (ORR) | assessed up to 1 year
  the proportion of patients with complete response and partial response , using RECIST v 1.1

SECONDARY OUTCOMES:
3-year disease free survival (3yr-DFS) | assessed up to 3 year
  the percentage of Primary thymoma patients without recurrence/metastasis within 3 years in all enrolled patients
overall survival rate (OS) | assessed up to 3 year
  from date of enrolment to date of death of any reason
Incidence of adverse events | assessed up to 1 year
Surgical conversion success rate | assessed up to 1 year
  Following chemotherapy to evaluate proportion of patients underwent timely operation
Pathologic Complete Response（pCR） | assessed up to 1 year
  the proportion of patients with complete response , using RECIST v 1.1
Main pathological Response | assessed up to 1 year
  the proportion of patients with complete response and partial response , using RECIST v 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Yian Zhang, Shanghai, Shanghai Municipality, China